CLINICAL TRIAL: NCT02153086
Title: Rozerem 8 mg Tablets Specified Drug-use Survey: <Long-term Survey on Insomnia Associated With Sleep-onset Difficulty > - Transitional Survey From the Preceding Drug-use Survey -
Brief Title: Ramelteon 8 mg Tablets Specified Drug-use Survey: <Long-term Survey on Insomnia Accompanied by Difficulty Falling Asleep> - Transitional Survey From the Preceding Drug-use Survey -
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 293-011
Record Dates: First submitted 2014-05-29; First posted 2014-06-02 (Estimated); Results first posted 2016-10-13 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-08

CONDITIONS: Insomnia
Keywords: Pharmacological therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — ramelteon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ramelteon 8 mg Tablets
  Interventions: Drug: Ramelteon

INTERVENTIONS:
Drug: Ramelteon — Ramelteon tablets 8 mg
  Other Names: Rozerem 8 mg Tablets

SUMMARY:
The purpose of this survey is to examine the safety and efficacy of long-term use of ramelteon tablets (Rozerem 8 mg Tablets) in participants with difficulty falling asleep associated with insomnia in daily medical practice.

DETAILED DESCRIPTION:
This survey was designed to examine the safety and efficacy of long-term use of ramelteon tablets (Rozerem 8 mg Tablets) in participants with difficulty falling asleep associated with insomnia in daily medical practice.The usual dosage for adults is 8 mg of ramelteon administered orally once daily at bedtime.

ELIGIBILITY:
Inclusion Criteria:

-Participants with difficulty falling asleep associated with insomnia who have completed a 4-week follow-up in the preceding drug use surveillance and are able to receive continuous administration of Rozerem Tablets

Exclusion Criteria:

* Participants with contraindications to Rozerem Tablets.
* Participants with previous history of hypersensitivity to ingredients in Rozerem Tablets.
* Participants with severe liver dysfunction.
* Participants taking fluvoxamine maleate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Insomnia
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2011-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Postmarketing Group Manager, Study Chair — Takeda
Locations (2):
- Japan (2):
  - Osaka
  - Tokyo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in Japan from 01 March 2011 to 30 June 2014.
Pre-assignment Details: Participants with a historical diagnosis of insomnia which was associated with difficulty in falling asleep in daily clinical practice were enrolled in a single treatment group to receive ramelteon 8 milligram (mg).
Groups:
- Ramelteon 8 mg: Participants receiving ramelteon 8 mg, tablet, orally, once as daily clinical practice were observed for up to 6 months. A follow up of 6 months was carried out.
Period: Overall Study
Arm/Group | Ramelteon 8 mg
Started | 236
Completed | 232
Not Completed | 4
Not completed — Not enrolled >=28 days and <=56 days | 2
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Population: The safety analysis set was defined as all participants who were enrolled and completed the study.
Arm/Group | Ramelteon 8 mg
Number analyzed (Participants) | 232
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (18.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 139
  Male | 93
Type of sleep disorders (Major symptoms) [Number; unit: participants] — Type of sleep disorders were classified on the basis of major symptoms as difficulty falling asleep, difficulty getting sound sleep, difficulty staying asleep, early morning awakening, and unknown.
  participants
    Difficulty falling asleep | 127
    Difficulty getting sound sleep | 16
    Difficulty staying asleep | 44
    Early morning awakening | 2
    Unknown | 43
Degree of sleep disorders [Number; unit: participants] — Degree of sleep disorders were categorized on the basis of severity, as mild, moderate or severe.
  participants
    Mild | 72
    Moderate | 130
    Severe | 30
Duration of insomnia [Number; unit: participants]
  Less than (<) 1 year | 102 (2.71)
  Greater than equal to (>=) 1 year to <3 years | 15
  >=3 to <5 years | 14
  >=5 years | 11
  Unknown | 90
Presence of complications [Number; unit: participants]
  Had Complications | 193
  Had No Complications | 39
Breakdown of complications [Number; unit: participants] — Complications were categorized as hypertension, dyslipidaemia, mental disease, allergic disease, diabetes mellitus, heart or cerebrovascular disease, and renal and urinary disorders. Participants may be represented in more than 1 category.
  participants
    Hypertension | 86
    Dyslipidaemia | 57
    Mental disease | 32
    Allergic disease | 23
    Diabetes mellitus | 22
    Heart or cerebrovascular disease | 22
    Renal and urinary disorders | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting One or More Adverse Drug Reactions
Description: Adverse drug reactions are defined as adverse events (AEs) which are in the investigator's opinion of causal relationship to the study treatment. AEs are defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product reported from the first dose of study drug to the last dose of study drug.
Time Frame: Baseline up to 12 months
Population: The safety analysis set was defined as all participants who were enrolled and completed the study.
Measure: Number; unit: participants
Arm/Group | Ramelteon 8 mg
Number analyzed (Participants) | 232
participants | 0

2. Secondary Outcome: Sleep Status: Sleep Onset Latency
Description: Sleep status was determined by measuring the sleep onset latency, defined as the length of time taken from lying down for the night until sleep onset. The data was assessed at baseline, Week 4 and final visit (last visit for a participant in the study, up to Month 12).
Time Frame: Baseline, Week 4 and Month 12
Population: The efficacy assessment population was defined as participants whose efficacy data at baseline and at least 1 post-baseline time points was available.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ramelteon 8 mg
Number analyzed (Participants) | 207
minutes
  Baseline (n=143) | 98.7 (73.3)
  At Week 4 (n=109) | 48.3 (57.6)
  At Final Assessment (n=127) | 38.9 (39.4)

3. Secondary Outcome: Sleep Status: Total Sleep Time
Description: Sleep status was determined by measuring the total sleep time, defined as the amount of actual sleep time during a sleep episode. The data was assessed at baseline, Week 4 and final visit (last visit for a participant in the study, up to Month 12).
Time Frame: Baseline, Week 4 and Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ramelteon 8 mg
Number analyzed (Participants) | 207
hours
  Baseline (n=137) | 6.74 (2.11)
  At Week 4 (n=102) | 7.51 (1.64)
  At Final Assessment (n=120) | 7.46 (1.72)

4. Secondary Outcome: Sleep Status: Number of Awakenings
Description: Sleep status of participants was assessed and summarized by calculating the number of times participants had awaken from the time of start of the investigation. The data was assessed at baseline, Week 4 and final visit (last visit for a participant in the study, up to Month 12).
Time Frame: Baseline, Week 4 and Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: number of awakenings
Arm/Group | Ramelteon 8 mg
Number analyzed (Participants) | 207
number of awakenings
  Baseline (n=150) | 2.3 (1.5)
  At Week 4 (n=115) | 1.2 (1.2)
  At Final Assessment (n=136) | 1.1 (1.1)

5. Secondary Outcome: Percentage of Participants Reported With Improvement on the Patient Global Impression (PGI) Scale for Sleep Onset
Description: Sleep onset was defined as the transition from wakefulness into sleep. PGI is a participant rated instrument to measure participant's change in overall status on a 7-point scale. Participants provide their response on a PGI questionnaire. Total score range from 1 (very much improved) to 7 (very much worse). Percentage of participants with improvement rated as "much better" or "a little better" were reported. The data was assessed at Week 4, Week 52 and final visit (follow up visit up to Month 12).
Time Frame: At Week 4, 52, and final assessment (up to 12 months)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Ramelteon 8 mg
Number analyzed (Participants) | 207
percentage of participants
  At Week 4 (n=207) | 80.2 (1.5)
  At Week 52 (n=88) | 93.2 (1.2)
  At Final Assessment (n=207) | 85.5 (1.1)

6. Secondary Outcome: Percentage of Participants Reported With Improvement on the PGI Scale for Sleep Duration
Description: Sleep duration was defined as the total amount of sleep obtained. PGI is a participant rated instrument to measure participant's change in overall status on a 7-point scale. Participants provide their response on a PGI questionnaire. Total score range from 1 (very much improved) to 7 (very much worse). Percentage of participants with improvement rated as "much better" or "a little better" were reported. The data was assessed at Week 4, Week 52 and final visit (follow up visit up to Month 12).
Time Frame: At Week 4, 52, and final assessment (up to 12 months)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Ramelteon 8 mg
Number analyzed (Participants) | 207
percentage of participants
  At Week 4 (n=207) | 77.8 (1.5)
  At Week 52 (n=88) | 93.2 (1.2)
  At Final Assessment (n=207) | 84.0 (1.1)

7. Secondary Outcome: Percentage of Participants Reported With Improvement on the PGI Scale for Sleep Quality
Description: Sleep quality was defined as participants satisfaction of the sleep experience, integrating aspects of sleep initiation, sleep maintenance, sleep quantity, and refreshment upon awakening. PGI is a participant rated instrument to measure participant's change in overall status on a 7-point scale. Participants provide their response on a PGI questionnaire. Total score range from 1 (very much improved) to 7 (very much worse). Percentage of participants with improvement rated as "much better" or "a little better" were reported. The data was assessed at Week 4, Week 52 and final visit (follow up visit up to Month 12).
Time Frame: At Week 4, 52, and final assessment (up to 12 months)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Ramelteon 8 mg
Number analyzed (Participants) | 207
percentage of participants
  At Week 4 (n=207) | 80.2 (1.5)
  At Week 52 (n=88) | 93.2 (1.2)
  At Final Assessment (n=207) | 86.0 (1.1)

8. Secondary Outcome: Percentage of Participants Reported With Improvement on the PGI Scale for Morning Awakening
Description: Morning awakening was defined as the return to the awaked state from any non-rapid eye movement (NREM) to rapid eye movement (REM) sleep stages in the morning. PGI is a participant rated instrument to measure participant's change in overall status on a 7-point scale. Participants provide their response on a PGI questionnaire. Total score range from 1 (very much improved) to 7 (very much worse). Percentage of participants with improvement rated as "much better" or "a little better" were reported. The data was assessed at Week 4, Week 52 and final visit (follow up visit up to Month 12).
Time Frame: At Week 4, 52, and final assessment (up to 12 months)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Ramelteon 8 mg
Number analyzed (Participants) | 207
percentage of participants
  At Week 4 (n=207) | 67.6 (1.5)
  At Week 52 (n=88) | 87.5 (1.2)
  At Final Assessment (n=207) | 77.8 (1.1)

9. Secondary Outcome: Percentage of Participants Reported With Improvement on the PGI Scale for Remaining Tiredness in the Morning
Description: Remaining tiredness in the morning was defined as an experience of fatigue after complete or adequate sleep duration. PGI is a participant rated instrument to measure participant's change in overall status on a 7-point scale. Participants provide their response on a PGI questionnaire. Total score range from 1 (very much improved) to 7 (very much worse). Percentage of participants with improvement rated as "much better" or "a little better" were reported. The data was assessed at Week 4, Week 52 and final visit (follow up visit up to Month 12).
Time Frame: At Week 4, 52, and final assessment (up to 12 months)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Ramelteon 8 mg
Number analyzed (Participants) | 207
percentage of participants
  At Week 4 (n=207) | 72.5 (1.5)
  At Week 52 (n=88) | 81.8 (1.2)
  At Final Assessment (n=207) | 77.3 (1.1)

10. Secondary Outcome: Percentage of Participants Reported With Improvement on the PGI Scale for Daytime Somnolence
Description: Daytime somnolence was defined as excessive daytime sleepiness (EDS), characterized by general lack of energy, even after adequate or prolonged night time sleep. PGI is a participant rated instrument to measure participant's change in overall status on a 7-point scale. Participants provide their response on a PGI questionnaire. Total score range from 1 (very much improved) to 7 (very much worse). Percentage of participants with improvement rated as "much better" or "a little better" were reported. The data was assessed at Week 4, Week 52 and final visit (follow up visit up to Month 12).
Time Frame: At Week 4, 52, and final assessment (up to 12 months)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Ramelteon 8 mg
Number analyzed (Participants) | 207
percentage of participants
  At Week 4 (n=207) | 65.2 (1.5)
  At Week 52 (n=88) | 81.8 (1.2)
  At Final Assessment (n=207) | 76.8 (1.1)

11. Secondary Outcome: Percentage of Participants Reported With Improvement on the PGI Scale for Daytime Physical Condition/Function
Description: Daytime physical condition/function was defined as general condition of participant throughout the day after adequate or prolonged night time sleep. PGI is a participant rated instrument to measure participant's change in overall status on a 7-point scale. Participants provide their response on a PGI questionnaire. Total score range from 1 (very much improved) to 7 (very much worse). Percentage of participants with improvement rated as "much better" or "a little better" were reported. The data was assessed at Week 4, Week 52 and final visit (follow up visit up to Month 12).
Time Frame: At Week 4, 52, and final assessment (up to 12 months)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Ramelteon 8 mg
Number analyzed (Participants) | 207
percentage of participants
  At Week 4 (n=207) | 70.5 (1.5)
  At Week 52 (n=88) | 84.1 (1.2)
  At Final Assessment (n=207) | 77.3 (1.1)

ADVERSE EVENTS:
Time Frame: Baseline up to 12 months
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Only adverse drug reactions were analyzed in this study.
Arm/Group | Ramelteon 8 mg
Serious Adverse Events (participants affected / at risk) | 0/232
Other Adverse Events (participants affected / at risk) | 0/232

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.